CLINICAL TRIAL: NCT04737291
Title: Outcomes of Drug Coated Balloon Angioplasty for Femoropopliteal Lesions in Patients With Critical Limb Ischemia
Brief Title: Drug Coated Ballon in Critical Limb Ischemia
Acronym: DCB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Nageeb, doctor, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: drug coated balloon
Record Dates: First submitted 2021-01-13; First posted 2021-02-03 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Drug Coated Balloon

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Angioplasty by DCB (Experimental): angioplasty of stenotic , ocluded or recoil segment using drug coated ballon
  Interventions: Device: drug coated balloon

INTERVENTIONS:
Device: drug coated balloon — use of drug coated balloon in treatment of critical limb ischemia

SUMMARY:
Evaluate the safety and efficacy of drug coated balloon (DCB) for the treatment of femoropopliteal lesions in patients with critical limb ischemia (CLI)

DETAILED DESCRIPTION:
Critical limb ischemia (CLI) is the most advanced stage of peripheral artery disease (PAD); which is estimated to affect more than 200 million people worldwide.(1) CLI classified as Rutherford category (RC) 4-6, includes ischemic rest pain and tissue loss.(2) The first line revascularization strategy for patients with CLI is endovascular percutaneous transluminal angioplasty (PTA).(3) The treatment of femoropopliteal lesions displays a huge anatomic challenge as this segment serves various biomechanical functions, Which makes endovascular treatment is challenging.(4) Plain balloon (PB) angioplasty for femoropopliteal artery disease has a high rate of procedural success and an acceptable safety profile, in spite of initially encouraging technical success after femoropopliteal (PTA), postprocedural restenosis remains the major challenge(5) Excessive extracellular matrix material synthesized by activated smooth muscle cells (SMC) in the media of the arteries leads to Neointimal hyperplasia and restenosis.(6) Restenosis resulting in loss of primary patency, late lumen loss (LLL), occlusion and/or the need for target lesion revascularization (TLR).(7) Drug-coated balloons (DCBs) inhibit the neointimal hyperplasia, the biological mechanism of restenosis formation, by application of cytostatic agents in a local therapeutic concentration.(8) The antiproliferative paclitaxel (PTX) seems to be the most effective therapeutic agent for DCBs due to local retention in the arterial wall.(9)

ELIGIBILITY:
Inclusion criteria:

* Adults at least 18 years of age with critical lower limb ischemia (Rutherford category 4, 5), stenotic (≥70% by visual angiographic assessment) or occlusive lesions in the native SFA or PPA, and vessel diameter ≥4 and ≤6 mm were eligible.
* Total lesion length ≤190 mm (visual angiographic assessment).
* DE novo angioplasty
* Recurrent or recoil lesion

Exclusion criteria:

* pregnancy
* breast feeding
* iliac lesions
* Malignancy
* Patients with raised renal chemistry.
* Patients with contraindication to antiplatelet therapy.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-03-15 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Freedom from device- and procedure-related mortality | 30 days
  mortality related to procedure
30 days clinically driven target vessel revascularization | 30 days
  patency rate

SECONDARY OUTCOMES:
Major adverse events | 12 months
  major adverse events as amputation
1 year clinically driven target vessel revascularization | 12 months
  patency rate

CONTACTS AND LOCATIONS:
Overall Officials: hassan bakr, professor, Study Chair — Assiut University; mahmoud ismael, ass profesor, Study Director — Assiut University; osman mahmoud, lecturer, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided